CLINICAL TRIAL: NCT04747574
Title: A Phase I Feasibility Study to Evaluate the Safety of CD24-Exosomes in Patients With Moderate/Severe COVID-19 Infection
Brief Title: Evaluation of the Safety of CD24-Exosomes in Patients With COVID-19 Infection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Eli Sprecher, MD, Nadir Arber MD, MSc, MHA Professor of Medicine and Gastroenterology. Head of the Health Promotion Center and the Integrated Cancer Prevention Center Tel-Aviv Sourasky Medical Center, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0254-20-TLV
Record Dates: First submitted 2021-01-26; First posted 2021-02-10 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: SARS-CoV-2
Keywords: SARS-CoV-2; Severe acute respiratory syndrome coronavirus 2; COVID-19; Exosomes; ARDS; CD24; CD-24 exosomes
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EXO-CD24 exosome treatment (Other): Group 1, 5 patients are treated with 1x10^8 exosome particles per 2 ml saline.
  Group 2: 5 patients are treated with 5x10^8 exosome particles per 2 ml saline.
  Group 3: 20 patients are treated with 1x10^9 exosomes particles per 2 ml saline.
  Group 4: 5 patients are treated with 1x10^10 exosomes particles per 2 ml saline.
  The drug is aerosolized in normal saline for inhalation and administered via a standard hospital-grade inhalation device, QD for 5 days. Study treatment is given as an add-on to the standard of care.
  Interventions: Drug: EXO-CD24

INTERVENTIONS:
Drug: EXO-CD24 — The study active treatment is EXO-CD24 -exosomes (natural nano-sized vesicles secreted by human cells) that were engineered to overexpress CD24, aerosolized in normal saline for inhalation via a standard hospital-grade inhalation device, QD for 5 days.

SUMMARY:
This is an open-label Phase I study, four dose escalation groups, to evaluate the safety of CD24-exosomes in patients with moderate/severe COVID-19 disease.

Patients with moderate/severe COVID-19 infection and factors predictive of a cytokine storm are recruited from the Corona department of the Tel Aviv Sourasky Medical Center (TASMC), who have provided informed consent are being recruited in four dose groups who will receive the exosome treatment as an add-on treatment to standard treatment.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is a highly transmissible disease in the community. The main cause of clinical deterioration that leads to death is the cytokine storm in the lung.

CD24 is a small heavily glycosylated GPI-anchored protein. CD24 is a key player in the vast majority of human cancers and also plays an important role in controlling the homeostatic proliferation of T cells. Hence, CD24 can negatively regulate inflammation.

The treatment is a biologic therapeutic agent based on exosomes carrying CD24. The rationale for this treatment is that exosomes overexpressing CD24, isolated and purified from T-REx™-293 cells engineered to express CD24 at high levels, can suppress the cytokine storm and are delivered directly to the target organ using exosomes as a highly body-compatible delivery vehicle. This enables a strong reduction of the required dose (as opposed to systemic administration), and reduces the risk for adverse events.

ELIGIBILITY:
1. A COVID-19 diagnosis confirmed with a SARS-CoV-2 viral infection positive polymerase chain reaction (PCR) test
2. Disease severity: Moderate/severe according to the following criteria (at least one clinical parameter and one laboratory parameter are required):

   1. Clinical and Imaging-based evaluation

      * Respiratory rate > 23/ min and < 30/min
      * SpO2 at room air ≤94% and ≥90%
      * Bilateral pulmonary infiltrates >50% within 24-48 hours or a severe deterioration compared to imaging at admission
   2. Evidence of an exacerbated inflammatory process

      * LDH score > 450 u/L
      * CRP >100 u/L
      * Ferritin >1650 ng/ml
      * Lymphopenia <800 cells/mm3 v. D-dimers>1
3. Willing and able to sign an informed consent

Exclusion Criteria:

1. Age<18 years or >85 years
2. Any concomitant illness that, based on the judgment of the Investigator is terminal
3. Ventilated patient
4. Pregnancy (positive urine pregnancy test [women of childbearing potential only]) or breastfeeding
5. Unwilling or unable to provide informed consent
6. Participation in any other study in the last 30 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-02-25 (Estimated); Study Completion 2021-03-25 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint: Adverse events | 35 days
  Number of adverse events, and adverse events leading to premature study termination.

SECONDARY OUTCOMES:
Exploratory Endpoint: Alive at Day 5 without bronchospasms, unexpected infections, or clinical deterioration | 5 days
  A composite endpoint comprised of alive at Day 5 without bronchospasms, unexpected infections, or a significant clinical deterioration compared to Baseline
Exploratory Endpoint: Proportion of patients with respiratory rate ≤ 23/min for 24 hours | 5 days
  Proportion of patients with respiratory rate ≤ 23/min for 24 hours
Exploratory endpoint: Change in respiratory rate from baseline to Day 5 | 5 days
  Change in respiratory rate from baseline to Day 5
Exploratory endpoint: Proportion of patients with SpO2 saturation ≥94% for at least 24 hours | 5 days
  Proportion of patients with SpO2 saturation ≥94% for at least 24 hours
Exploratory endpoint: Change in SpO2 saturation from baseline to Day 5 | 5 days
  Change in SpO2 saturation from baseline to Day 5
Exploratory endpoint: Proportion of patients with no artificial ventilation after 5 days of treatment | 5 days
  Proportion of patients with no artificial ventilation after 5 days of treatment
Exploratory endpoint: Proportion of patients with a change in absolute lymphocyte count, sustained for ≥48 hours after 5 days of treatment | 7 days
  Proportion of patients with a change in the absolute lymphocyte count, sustained for ≥48 hours after 5 days of treatment
Exploratory endpoint: Change in the absolute lymphocyte count from baseline to Day 5 | 5 days
  Change in the absolute lymphocyte count from baseline to Day 5
Exploratory endpoint: Change in neutrophil-to-lymphocyte ratio (NLR), sustained for ≥48 hours after 5 days of treatment | 7 days
  Proportion of patients with a change in the neutrophil-to-lymphocyte ratio, sustained for ≥48 hours after 5 days of treatment
Exploratory endpoint: Change in neutrophil-to-lymphocyte ratio (NLR) from baseline to Day 5 | 5 days
  Change in neutrophil-to-lymphocyte ratio (NLR) from baseline to Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Nadir Arber, Prof., Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No